CLINICAL TRIAL: NCT02693275
Title: Reference Database Development for the Quotient® System iPad Test (Ages 6 - 80 Years Old)
Brief Title: Reference Database Development for the Quotient® System iPad Test
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pearson/Clinical Assessment (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: PNB&I-4001
Record Dates: First submitted 2016-02-23; First posted 2016-02-26 (Estimated); Last update posted 2017-04-05 (Actual); Status verified 2017-04

CONDITIONS: Healthy Volunteers
Keywords: Community Sampling

STUDY DESIGN:
Masking Description: Open Label
Oversight: Data Monitoring Committee: No

ARMS (1):
- Quotient® System iPad Test (Other): The Quotient® System iPad Test is a test specifically designed to provide clinicians with objective measures in ability to maintain seated stillness, sustained attention to a monotonous task and inhibiting incorrect impulsive responses. The attention task with motion analyses provides a number of objective measures for detailed assessment of the subject's movements and attentiveness.
  Interventions: Device: Quotient® System iPad Test

INTERVENTIONS:
Device: Quotient® System iPad Test — See arm/group description
  Other Names: Quotient®

SUMMARY:
This study is being conducted to create a database for the Quotient® System iPad Test. Using community sampling, NCS Pearson will compile the results of this study to create a database against which the results of clinical Quotient tests may be compared to determine patient performance relative to the expected results for developmental age and gender.

DETAILED DESCRIPTION:
Study Design:

This study is being conducted at 4 clinical sites and consists of up to two study visits. All study participants will complete at least one study visit. A smaller cohort of participants will complete a second visit for the purpose of assessing test retest reliability across the study sample. Subjects will be recruited using the clinic's relevant patient population and IRB approved recruitment material. Interested volunteers will participate in an initial screening, which may be done by telephone or in person that will be conducted by the clinic's research staff. Upon preliminary confirmation that the subject meets all inclusion criteria and does not meet any exclusion criteria, an appointment will be scheduled for the first study visit.

At the first visit, the study will be explained in detail. Adults will be asked to provide written informed consent. Parents or guardians of individuals under the age of 18 years old will provide written informed consent on behalf of the minor. Individuals between the age of 7 and 18 years of age will also provide their written assent. All consents and assents will be obtained prior to any study procedure being performed. Following consent, a brief medical history, including current medications the subject is taking, will be obtained. Subjects will complete a standard self-assessment questionnaire, appropriate for age, to screen for presence of ADHD. Subjects will not be excluded from the study based on responses to the questionnaire but their results will be considered in the analysis of study data. All subjects will take the appropriate version; Child (ages 6 -12.11), Adolescent (ages 13 - 19.11), or Adult (ages 20 - 79.11) of the 15-minute Quotient® System iPad Test.

At this visit, a cohort of participants across 7 age groups will be asked to return the clinic for a second study visit. These participants will be asked, in consecutive order of enrollment, to return to the clinic for a second study visit. Study participants who complete visit one are not required to participate in the retest cohort group and may opt out of returning to the clinic for visit two. Once the required number of participants (350 - 400) have completed the second study visit, that portion of the study will be closed to further enrollment and no further subjects will be given the option to return for the retest visit (visit 2).

Retest Visit 2 will occur 7 - 14 days following study visit 1. Subjects will be assessed for changes in health status and current medications since the time of visit 1. Subjects will repeat the appropriate version (Child, Adolescent or Adult) of the 15-minute Quotient® System iPad Test.

● Study Enrollment: A minimum of 1440 subjects with oversampling of 11%. Total enrollment is expected to be approximately 1600.

● Study Population:

Visit 1:

Male and female subjects from the age of 6 years until the age of 80 years. There will be a total of 16 age bands with approximately 90 subjects enrolled in each age band. Optimally, there will be a 50-50-male/female-gender stratification per each age category.

Visit 2:

A cohort of at least 350 subjects who have completed study Visit 1 will be asked to return for Visit 2. An oversampling of 11% is anticipated bringing the total number of subjects asked to return for Visit 2 to approximately 400. Visit 2 will include both male and female participants from 7 age bands.

* Study Procedures:

  1. Review Inclusion/Exclusion Criteria
  2. Obtain Written Adult Informed Consent
  3. Obtain Written Minor Informed Assent
  4. Verbal Report of Medical History
  5. Concomitant Medications
  6. Self-assessment Questionnaire:

     1. ADHD Self Rating Scale (ADHDRS-IV) for subjects ages 6 - 19.11
     2. ADHD Symptom Rating Scale (ASRS-V1.1) for subjects ages 20 - 79.11
  7. Quotient® System iPad Test - Child, Adolescent or Adult test as appropriate for age
* Study Duration:

Dependent on accrual but estimated to be six (6) months to nine (9) months.

● Statistical Analysis Plan: The data of the study will be used to identify normative ranges and percentiles by age and gender. Each age range group of 90 will be compared for group differences between genders, and evaluated for the effects of age on performance. The SPSS software (SPSS Inc., Chicago, Illinois) will be used for statistic procedures in this study.

ELIGIBILITY:
Inclusion Criteria:

1. Male or Female
2. Ages 6 years - 79 years and 11 months (79.11) of age
3. Report of good physical health
4. Able to understand test instructions and comply with testing
5. Willing to give written informed consent and/or assent

Exclusion Criteria:

1. History of known neurological disease or insult (e.g., head trauma with LOC, skull fracture, seizure disorders). History of febrile seizure does not exclude subject from study participation
2. Major Medical Disorders known to the Investigator that would make it difficult for the participant to complete study requirements
3. Any major medical or neurological condition that could affect motor activity or attention (e.g. Parkinson's, MS, dementia)
4. Currently ill with cold, flu or infections which may compromise their ability to perform the computer task
5. Any condition in which the investigator deems the subject inappropriate for participation in the study

Ages: 6 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 1333 (Actual)
Dates: Start 2016-04; Primary Completion 2017-03-31 (Actual); Study Completion 2017-03-31 (Actual)

PRIMARY OUTCOMES:
Range of measured head motion of typically developing subjects while taking the attention test as determined on the dimensions of total number of motions >1mm/sec during the 15-minute test | 12 Months
  The result of this primary outcome measure will be analyzed statistically to establish the range of measured values for this assessment parameter and the population distribution of the measurement in typically developing subjects stratified for age, gender and ethnicity.
Duration of motion free periods in seconds during the 15-minute test | 12 Months
  The result of this primary outcome measure will be analyzed statistically to establish the range of measured values for this assessment parameter and the population distribution of the measurement in typically developing subjects stratified for age, gender and ethnicity.
Area of head motion covered in centimeters during the total 15-minute test. | 12 Months
  The result of this primary outcome measure will be analyzed statistically to establish the range of measured values for this assessment parameter and the population distribution of the measurement in typically developing subjects stratified for age, gender and ethnicity.
Total length of movement in meters during the total 15-minute test. | 12 Months
  The result of this primary outcome measure will be analyzed statistically to establish the range of measured values for this assessment parameter and the population distribution of the measurement in typically developing subjects stratified for age, gender and ethnicity.
Range of attentive responses to a 15-minute go/no-go attention task (assessed simultaneously with the motion assessment) in terms of accuracy in % correct response during the 15-minute test | 12 Months
  The result of this primary outcome measure will be analyzed statistically to establish the range of measured values for this assessment parameter and the population distribution of the measurement in typically developing subjects stratified for age, gender and ethnicity.
Average response time to stimulus items in milliseconds during the 15-minute test | 12 Months
  The result of this primary outcome measure will be analyzed statistically to establish the range of measured values for this assessment parameter and the population distribution of the measurement in typically developing subjects stratified for age, gender and ethnicity.
Total errors of omission in % of total targets during the 15-minute test | 12 Months
  The result of this primary outcome measure will be analyzed statistically to establish the range of measured values for this assessment parameter and the population distribution of the measurement in typically developing subjects stratified for age, gender and ethnicity.
Total errors of commission in % of total non-targets during the 15-minute test | 12 Months
  The result of this primary outcome measure will be analyzed statistically to establish the range of measured values for this assessment parameter and the population distribution of the measurement in typically developing subjects stratified for age, gender and ethnicity.
Variability reported as the standard deviation of all responses from mean response time reported in milliseconds during the 15-minute test | 12 Months
  The result of this primary outcome measure will be analyzed statistically to establish the range of measured values for this assessment parameter and the population distribution of the measurement in typically developing subjects stratified for age, gender and ethnicity.

CONTACTS AND LOCATIONS:
Overall Officials: Calvin R Sumner, MD, Principal Investigator — Pearson/Clinical Assessment
Locations (4):
- United States (4):
  - Center for Psychiatry and Behavioral Medicine, Inc., Las Vegas, Nevada
  - Growing Child Pediatrics, PA, Raleigh, North Carolina
  - Erickson Research and Development, Clinton, Utah
  - Tanner Clinic, Layton, Utah

IPD SHARING:
Plan to Share IPD: No